CLINICAL TRIAL: NCT02257931
Title: Resistance Pattern of Gram-negative Bacteria Isolated From Blood From HSCT Recipients.
Brief Title: Gram-negative Bacteremia in HSCT Recipients
Acronym: GNB
Status: Completed | Type: Observational
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Responsible Party: Sponsor
Other Study IDs: 8414106
Record Dates: First submitted 2014-10-02; First posted 2014-10-07 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Allogeneic or Autologous HSCT
Keywords: infection; bacteria; gram-negative; HSCT; allogeneic; autologous; recipients, of all ages, for any indications
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HSCT recipient: Allogeneic or autologous HSCT recipients, of all ages, for any indications. From this group we take those with a gram-negative bacteremia within 6 months after HSCT.

SUMMARY:
A significant increase in resistant bacteria emerging in HSCT recipients. For example, 25% - 42% of all enterobacteriaceae produce extended spectrum beta-lactamases; 8 - 72% of Pseudomonas aeruginosa are resistant to at least one and 25 - 62% to three or more antibiotic classes, 13% of Gram-negative bacteria are caused by a multidrug-resistant (MDR) strain (Trecarichi JI 09, Mikulska BBMT 09, Oliveira BMT 07, Caselli Haemat 10, Gudiol, JAC 11). These resistant bacteria may be associated with increased mortality and have limited treatment options (Caselli Haemat 10, Poutsiaka BMT 07, DiazGranadoz JID 05). To provide the currently best empirical coverage and to control the growing resistance, knowledge of trends in antibiotic susceptibility, as well as risk factors is essential. For this reason we propose to perform non-interventional prospective multicentre study in EBMT centres.

DETAILED DESCRIPTION:
Primary objective:

To determine the incidence and pattern of antimicrobials resistance among Gram-negative bacteria isolated from blood in HSCT patients during the first 6 months after the transplantation.

Secondary Objective(s):

2) to determine whether the currently administered empirical therapy is appropriate; 3) to determine mortality associated with resistant vs. sensitive Gram-negative bacteria

Primary endpoints:

The proportion of resistant pathogens among gram-negative bacterial pathogens isolated from blood of HSCT recipients during the first 6 months post HSCT.

1. Pathogens resistant to either one of the following: ceftazidime or cefepime or piperacillin-tazobactam
2. Pathogens with carbapenem resistance (not including ertapenem)
3. MDR pathogens

Secondary endpoints:

1. The proportion of resistant Gram-negative pathogens not listed in the primary end-point among Gram-negative bacterial pathogens isolated from blood of HSCT recipients during the first 6 months post HSCT:

   * Gram-negative pathogens resistant to fluoroquinolones
   * Gram-negative pathogens resistant to at least one of aminoglycosides
   * Gram-negative pathogens resistant to colistin
   * Gram-negative pathogens (other than Pseudomonas) resistant to tigecycline
   * Acinetobacter spp. resistant to ampicillin-sulbactam
   * Acinetobacter spp. resistant to tetracyclin or minocycline
   * Stenotrophomonas maltophilia resistant to trimethoprim-sulfamethoxazole
   * Stenotrophomonas maltophilia resistant to minocycline
2. The outcome of the infections caused by resistant pathogens vs. sensitive, including mortality of any cause within 7 days and within 30 days;
3. The appropriateness of the currently administered empirical antimicrobial therapy; Inappropriate initial antimicrobial therapy will be defined as empirical antibiotic regimen, given in the first 48 hours following obtaining the blood cultures, that does not include at least one antibiotic that is active in vitro against the infecting microorganism.

Research design:

Data on all the episodes of Gram-negative bacteria blood stream infections will be collected prospectively from the initiation of the conditioning treatment until the end of the first 6 months after the HSCT (or death or lost follow-up, if they occur earlier).

Data on the patients who will develop Gram-negative infection will be reported using special MED C form and include data on the pathogen and antimicrobial susceptibility of the pathogen, treatment and outcome, and presence of certain risk factors, in addition to the data present in MED A form.

Patient's data such as age, gender, primary diagnosis and status of the disease, presence of co-morbidities, HSCT type, donor type, conditioning regimen (myeloablative versus reduced intensity), GVHD prophylaxis and outcome at the time of report will be obtained from the MED A form.

Study Population:

Inclusion criteria: Allogeneic or autologous HSCT recipients, of all ages, for any indications.

Exclusion criteria: Patients who are not willing to participate. Expected number of patients: 3650 HSCT patients to be recruited and followed in order to obtain data on 365 Gram negative episodes.

Basis for calculations:

Clinical assumptions

~30% of HSCT patients will have bacteremia, about a half of them due to Gram negatives=10-15% of HSCT patients. Depending on local epidemiology, about a 40% of them will be resistant to at least one of the antibiotics mentioned in the primary endpoint. Mortality in resistant GN bacteremia is 30-50%. Mortality in sensitive bacteremia is 5-20%.

Statistical issues

* The actual sample size for the analyses will be the number N* of episodes of Gram-negative bacteremia observed. These will be observed in N≤N* patients. For simplicity, we will assume that one patient ↔ one episode, i.e. N=N*.
* The total number of transplants that we should have in the participating centers during the recruitment period in order to observe N patients with (at least) an episode of Gram-negative bacteremia will be indicated by T. We will assume that N = 10% of T.
* Notice thus that these scenarios are "conservative", as we could expect to observe more patients with an episodes than 10%, and multiple episodes per patient.
* We considered several scenarios computing the minimum sample size necessary to obtain an estimation of the incidence of resistance among Gram-negative bacteremia episodes with precision equal to 0.05 (preferably) or 0.1, assuming a value between 20% and 60% for the incidence. (Confidence level for the interval estimate always equal to 95%). Scenarios have also been considered for secondary objectives. All calculations were done using the NCSS-PASS 2000 software.

T=365 transplants (N=3650 patients) is a minimum number of transplants necessary to be able to get a 95%CI=(0.35,0.45) when the actual incidence of resistance is equal to 40%.

Data Collection & Statistical Analysis Plan:

Center registration form will be sent to all EBMT centers before the beginning of the study. It will assess their willingness to participate and provide some background information on the number of transplants performed/year, names of the responsible persons, methods used by laboratories, etc. All episodes of blood stream Gram-negative bacterial infections will be collected prospectively since the initiation of the conditioning treatment and further on during the 6 months after the transplantation. All the episodes of Gram-negative bacteremias will be included, including multiple episodes in the same patient. For each episode of Gram-negative bacteremia, additional information including relevant microbiological data will be collected using MED C form. MED C form will include data on each Gram- negative isolate. Note, each time that the patient has a new positive blood culture for Gram - negative bacteria, a new MED C form should be filled. Repeated isolation of same pathogen, with same in vitro susceptibility will be considered as one isolate. We ask that MED C forms will be sent within 3 months from the end of the episode.

The baseline data on all the patients who will develop blood stream Gram-negative bacterial infections during the study period will be reported using the MED A form, which is routinely filled for all patients in the centers that belong to the EBMT. We ask that it will be filled within 3 months from the end of the 6 months after HSCT (or earlier if the patient ceased).

Resistance to antibiotics will be studied by in-vitro sensitivity tests performed by the local laboratories. The characteristics of the local laboratories, including essential data on methods used to determine susceptibility of isolates and guidelines used to determine susceptibility will be reported in the Centre Registration Form.

The collaborator from each center will be responsible for the reports from laboratories.

Statistical analysis The analysis of the data will be mostly descriptive. The incidence of resistance will be computed as a percentage, the denominator being the number of episodes of Gram-negative bacteremia, and the numerator being the number of episodes classified as "resistant". The relationship between Resistance and prognostic factors / characteristics will be investigated mostly in univariate analysis, applying standard summary measures (tables, quantiles) and non-parametric tests (chi-squared or Fisher Exact, Mann-Whitney or Kruskal-Wallis) - for categorical and continuous variables respectively. Possibly, a multivariate analysis could also be applied, using logistic regression; random effects models or GEE could be used to account for dependence of observations - nested by patient and center. The short-term mortality (at 7 and 30 days) will be computed as a percentage - unless a relevant proportion of loss to follow-up will be observed.

All data collection will be performed by the IDWP data office (Leiden) according to EBMT guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic or autologous HSCT recipients, of all ages, for any indications.

Exclusion Criteria:

* Patients who are not willing to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: eligible patients from EBMT centres
Sampling Method: Non-Probability Sample
Enrollment: 591 (Actual)
Dates: Start 2014-02; Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
The proportion of resistant pathogens among gram-negative bacterial pathogens isolated from blood of HSCT recipients during the first 6 months post HSCT. | 6 months after HSCT
  1. Pathogens resistant to either one of the following: ceftazidime or cefepime or piperacillin-tazobactam
  2. Pathogens with carbapenem resistance (not including ertapenem)
  3. MDR pathogens

SECONDARY OUTCOMES:
The proportion of resistant Gram-negative pathogens not listed in the primary end-point among Gram-negative bacterial pathogens isolated from blood of HSCT recipients during the first 6 months post HSCT: | 6 months after HSCT
  Gram-negative pathogens resistant to fluoroquinolones
  * Gram-negative pathogens resistant to at least one of aminoglycosides
  * Gram-negative pathogens resistant to colistin
  * Gram-negative pathogens (other than Pseudomonas) resistant to tigecyclin
  * Acinetobacter spp. resistant to ampicillin-sulbactam
  * Acinetobacter spp. resistant to tetracyclin or minocycline
  * Stenotrophomonas maltophilia resistant to trimethoprim-sulfamethoxazole
  * Stenotrophomonas maltophilia resistant to minocycline

OTHER OUTCOMES:
The outcome of the infections caused by resistant pathogens vs. sensitive, including mortality of any cause within 7 days and within 30 days; | 30 days after HSCT
The appropriateness of the currently administered empirical antimicrobial therapy | 6 months after HSCT
  The appropriateness of the currently administered empirical antimicrobial therapy; Inappropriate initial antimicrobial therapy will be defined as empirical antibiotic regimen, given in the first 48 hours following obtaining the blood cultures, that does not include at least one antibiotic that is active in vitro against the infecting microorganism.

CONTACTS AND LOCATIONS:
Overall Officials: Dina Averbuch, MD, Principal Investigator — Hadassah University Hospital, Pediatric Infectious Diseases Unit, Jerusalem, Israel; Dan Engelhard, MD, Principal Investigator — Hadassah University Hospital, Pediatric Infectious Diseases Unit, Jerusalem, Israel; Simone Cesaro, MD, Study Chair — Policlinico G.B. Rossi, paediatric haematology oncology, Verona, Italy
Locations (10):
- University Hospital Gasthuisberg, Leuven, Belgium
- First Affiliated Hospital of Soochow University, Suzhou, China
- University Hospital Center Rebro, Zagreb, Croatia
- Germany (2):
  - University of Muenster, Münster
  - Universitaetsklinikum Wuerzburg, Würzburg
- Rambam Medical Center, Haifa, Israel
- Inst. Portugues de Oncologia do Porto, Porto, Portugal
- Federal Research Centre for Pediatric Hematology, Moscow, Russia
- Karolinska University Hospital, Stockholm, Sweden
- Anadolu Medical Center, Kocaeli, Turkey (Türkiye)

REFERENCES:
- [Derived] Averbuch D, Tridello G, Hoek J, Mikulska M, Akan H, Yanez San Segundo L, Pabst T, Ozcelik T, Klyasova G, Donnini I, Wu D, Gulbas Z, Zuckerman T, Botelho de Sousa A, Beguin Y, Xhaard A, Bachy E, Ljungman P, de la Camara R, Rascon J, Ruiz Camps I, Vitek A, Patriarca F, Cudillo L, Vrhovac R, Shaw PJ, Wolfs T, O'Brien T, Avni B, Silling G, Al Sabty F, Graphakos S, Sankelo M, Sengeloev H, Pillai S, Matthes S, Melanthiou F, Iacobelli S, Styczynski J, Engelhard D, Cesaro S. Antimicrobial Resistance in Gram-Negative Rods Causing Bacteremia in Hematopoietic Stem Cell Transplant Recipients: Intercontinental Prospective Study of the Infectious Diseases Working Party of the European Bone Marrow Transplantation Group. Clin Infect Dis. 2017 Nov 13;65(11):1819-1828. doi: 10.1093/cid/cix646. PMID 29020364